CLINICAL TRIAL: NCT06935513
Title: Wearable Devices Empowering Active Health Initiatives for High-Risk Stroke Populations
Acronym: AISP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025005
Record Dates: First submitted 2025-03-30; First posted 2025-04-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Diabetes; Atrial Fibrillation; Dyslipidemia; Smoking; Physical Inactivity; Obesity and Overweight
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Atrial Fibrillation; Dyslipidemias; Smoking; Sedentary Behavior; Obesity; Overweight | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Wearable Devices (Experimental): Participants utilize wearable devices (smart wristbands) 24 hours a day for 6 months and receive medication reminders for each use and heart rate monitoring.
  Interventions: Behavioral: Wearable Devices
- Without Wearable Devices (No Intervention): Participants do not utilize wearable devices (smart wristbands) .

INTERVENTIONS:
Behavioral: Wearable Devices — Participants utilize wearable devices (smart wristbands) 24 hours a day for 6 months. Wearable devices can provide medication reminders for each use and heart rate monitoring.
  Arms: With Wearable Devices

SUMMARY:
The purpose of this study is to evaluate the control effect of smart wearable devices on key risk factors in the high-risk populations for stroke

DETAILED DESCRIPTION:
A randomized controlled study was conducted on the application of smart wearable devices in the intervention of high-risk populations for stroke, with a focus on whether the functions of smart wearable devices such as medication reminders, heart rate monitoring, and exercise reminders can effectively benefit the improvement of key risk factors for stroke, especially blood pressure, blood glucose, and blood lipids.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hypertension;
2. Diagnosed with diabetes;
3. Diagnosed with atrial fibrillation;
4. Smoking subjects;
5. Physical inactive subjects；
6. Obesity and overweight subjects;
7. Must be able to use smart wearable devices.

Exclusion Criteria:

1. Diagnosed with malignancies;
2. Diagnosed with psychiatric disorders;
3. Diagnosed with cognitive impairment;
4. Unable to operate smart wearable devices.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
medication adherence and risk factor control rates | 6 months
  1.The medication rates and control rates for hypertension; 2.The medication rates and control rates for hyperglycemia; 3. The medication rates and control rates for hyperlipidemia; 4.The medication rates and control rates for obesity.

SECONDARY OUTCOMES:
incident vascular events, including stroke, coronary heart disease (CHD), peripheral vascular disease (PVD), and other related cardiovascular events | 6 months
  Stroke is a sudden interruption of blood flow to the brain, caused by either a blockage (ischemic stroke) or rupture of a blood vessel (hemorrhagic stroke). Coronary heart disease is a cardiovascular condition characterized by the narrowing or blockage of the coronary arteries, the blood vessels that supply oxygen-rich blood to the heart muscle. Peripheral vascular diseases are circulatory disorders characterized by narrowing, blockage, or spasms in blood vessels outside the heart and brain, most commonly affecting arteries supplying the legs, arms, kidneys, or stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhong Ji, MD, PhD, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No